CLINICAL TRIAL: NCT00373867
Title: Behavioral Interventions for Low Back Pain
Brief Title: Effectiveness of Adding Behavioral Therapy to Physical Therapy to Treat Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R03AR051128 (NIH); R03AR051128 (NIH)
Record Dates: First submitted 2006-09-06; First posted 2006-09-08 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Low Back Pain
Keywords: Secondary prevention; Physical therapy; Fear-avoidance beliefs; Disability
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard (Active Comparator): Standard treatment-based classification physical therapy
  Interventions: Behavioral: Standard physical therapy
- Graded exercise (Active Comparator): Treatment-based classification physical therapy plus graded exercise
  Interventions: Behavioral: Graded exercise
- Graded exposure (Experimental): Treatment-based classification physical therapy plus graded exposure
  Interventions: Other: Graded exposure

INTERVENTIONS:
Behavioral: Standard physical therapy — Treatment-based classification physical therapy
  Arms: Standard
Behavioral: Graded exercise — Graded exercise increases an individual's tolerance to activity over time
  Arms: Graded exercise
Other: Graded exposure — Graded exposure places the individual in fearful situations and gradually increases their exposure to such situations.
  Arms: Graded exposure

SUMMARY:
Low back pain is a very common problem and the most common cause of job-related disability. While some occurrences of low back pain disappear within a couple of days, other occurrences take much longer to resolve or lead to more serious conditions. The purpose of this study is to determine the effectiveness of two behavioral types of therapy in reducing future disability in people who are receiving physical therapy for low back pain and tend to fear and avoid pain.

DETAILED DESCRIPTION:
Psychosocial factors, such as fear and avoidance, appear to play a role in the development of long-term disability from low back pain. The Fear-Avoidance Model of Exaggerated Pain Perception (FAMEPP) is a biopsychosocial model that attempts to explain how and why some individuals develop a more substantial psychological component to their low back pain problem than do others. FAMEPP suggests that an individual's pain-related fear and avoidance are the most important factors in determining whether long-term disability will result from an episode of low back pain. For example, FAMEPP suggests that individuals with high pain-related fear and avoidance are likely to use an avoidance response to low back pain, leading to both physical and psychological consequences. In contrast, individuals with low pain-related fear and avoidance are likely to use a confrontation type of response to low back pain and gradually return to their normal social and physical functioning.

Treatment based on FAMEPP involves two specific behavioral interventions that encourage people to confront their low back pain. The first intervention, graded exposure, places the individual in fearful situations and gradually increases their exposure to such situations. The second intervention, graded exercise, increases an individual's tolerance to activity over time. The purpose of this pilot study is to determine the effectiveness of graded exposure and graded exercise, when combined with traditional physical therapy, in reducing future disability in adults with low back pain who tend to fear and avoid pain.

Participants in this study will be randomly assigned to one of three groups:

* Group 1 will undergo graded exposure in addition to normal physical therapy during treatment sessions.
* Group 2 will undergo graded exercise in addition to normal physical therapy during treatment sessions.
* Group 3 will participate in only normal physical therapy during treatment sessions.

The number of treatment sessions will vary, depending on how a participant is improving. At Week 4 and Month 6, all participants will be evaluated with a pain symptom assessment and questionnaires on pain intensity, pain-related disability, fear-avoidance beliefs, overreaction to pain, and physical impairment. There will be no other follow-up visits for this study.

ELIGIBILITY:
Inclusion Criteria:

* Quebec Task Force Spinal Disorders (QTFSD) classification of 1a: acute low back pain without pain radiation below the gluteal fold
* QTFSD classification of 1b and 1c: subacute and chronic low back pain without pain radiation below the gluteal fold
* QTFSD classification of 2a: acute low back pain with pain radiation to the knee
* QTFSD classification of 2b and 2c: subacute and chronic low back pain with pain radiation to the knee
* QTFSD classification of 3a, 3b, or 3c: acute, subacute, or chronic low back pain with pain radiation below the knee
* Can read and speak English
* Parent or guardian willing to provide informed consent if applicable

Exclusion Criteria:

* QTFSD classification of 4a, 4b, or 4c: acute, subacute, or chronic low back pain with pain radiation below the knee and experiencing neurological symptoms
* QTFSD classification of 5: likely lumbar nerve root compression
* QTFSD classification of 6: confirmed lumbar nerve root compression
* QTFSD classification of 7: confirmed lumbar spinal stenosis
* QTFSD classification of 8: less than 6 months after surgery for back pain
* QTFSD classification of 9.1: more than 6 months after surgery for back pain and not experiencing any symptoms
* QTFSD classification of 11: other spinal disorders including cancer, disease inside bone, or fracture

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 108 (Actual)
Dates: Start 2006-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Measured at Week 4 and Month 6
Pain-related disability | Measured at Week 4 and Month 6

SECONDARY OUTCOMES:
Fear-avoidance beliefs | Measured at Week 4 and Month 6
Pain catastrophizing | Measured at Week 4 and Month 6
Physical impairment | Measured at Week 4 and Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Steven Z. George, PT, PhD, Principal Investigator — University of Florida
Locations (1):
- Shands Rehabilitation at the University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Result] George SZ, Zeppieri G Jr, Cere AL, Cere MR, Borut MS, Hodges MJ, Reed DM, Valencia C, Robinson ME. A randomized trial of behavioral physical therapy interventions for acute and sub-acute low back pain (NCT00373867). Pain. 2008 Nov 15;140(1):145-157. doi: 10.1016/j.pain.2008.07.029. Epub 2008 Sep 10. PMID 18786762
- [Result] Hirsh AT, George SZ, Bialosky JE, Robinson ME. Fear of pain, pain catastrophizing, and acute pain perception: relative prediction and timing of assessment. J Pain. 2008 Sep;9(9):806-12. doi: 10.1016/j.jpain.2008.03.012. Epub 2008 May 16. PMID 18486557
- [Result] George SZ, Fritz JM, Childs JD. Investigation of elevated fear-avoidance beliefs for patients with low back pain: a secondary analysis involving patients enrolled in physical therapy clinical trials. J Orthop Sports Phys Ther. 2008 Feb;38(2):50-8. doi: 10.2519/jospt.2008.2647. Epub 2008 Jan 22. PMID 18349490